CLINICAL TRIAL: NCT05728359
Title: Prospective Observational Study Investigating Genomic Determinants of Outcome From Cardiogenic Shock (GOlDilOCS)
Brief Title: Genomic Determinants of Outcome in Cardiogenic Shock
Acronym: Goldilocs
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 290406
Record Dates: First submitted 2022-09-22; First posted 2023-02-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiogenic Shock
Keywords: ACS,; Cardiogenic Shock; ECMO; Impella; Gene Expression; Endotype
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — We will collect blood samples (18ml per time-point) at research-specific time points Plasma will be extracted from spun blood in appropriate blood collection tubes (EDTA, 2x3mL), aliquoted and stored at -80°C.
  DNA will be extracted from the Buffy Layer of spun whole human blood. RNA from human whole blood (1x3ml) will be collected into a Tempus tube. Whole blood will be added to Cytodelics to allow cellular fixation and subsequent analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cardiogenic shock and MI: Patients presenting with acute myocardial infarction and cardiogenic shock who are supported medically (ie. inotropes +/- intra aortic balloon pump only). N=50
  Interventions: Other: Observational study
- Cardiogenic shock and MI wtih ECMO: Patients presenting with acute myocardial infarction and cardiogenic shock who are supported medically with ECMO (+/- LV unloading device). N=50
  Interventions: Other: Observational study
- Cardiogenic shock and MI wtih Impella: Patients presenting with acute myocardial infarction and cardiogenic shock who are supported medically with Impella. N=50
  Interventions: Other: Observational study
- MI without cardiogenic shock: Patients presenting with acute myocardial infarction and cardiogenic shock as a control comparator
  Interventions: Other: Observational study
- Non ischemic Cardiogenic Shock ie myocarditis: Patients presenting with myocarditis and cardiogenic shock as a control comparator
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Blood sampling and clinical data collection

SUMMARY:
The aim of this project is to understand the heterogeneity of both the immune consequences and treatment responses in CS. We will explore this heterogeneity through identification of transcriptomic sub-phenotypes and their association with outcomes, including therapeutic responses.

DETAILED DESCRIPTION:
This is a prospective observational cohort study in 8-10 cardiac centres across Europe. We will recruit patients presenting with acute myocardial infarction (AMI) and CS who are supported medically (n=100); with extracorporeal membrane oxygenation (n=50); and with the Impella Device (n=50). We will also enrol patients who present with either AMI and no evidence of CS (n=50) or CS due to non-ischaemic pathologies (e.g. myocarditis: n=50) as comparators. The recruitment target is 300 patients.

ELIGIBILITY:
Inclusion Criteria:

* All of the following are required for inclusion following screening:

  * Willing to provide informed consent or appropriate consent from a nominated consultee or personal consultee
  * Presentation within 24 hours of onset of ACS symptoms.
  * CS can only be secondary to ACS (Type 1 MI STEMI or N-STEMI) or myocarditis
  * Planned or completed revascularisation of culprit coronary artery

CS will be defined by:

* Systolic blood pressure <90 mmHg for at least 30 minutes
* A requirement for a continuous infusion of vasopressor or inotropic therapy to maintain systolic blood pressure > 90 mmHg.
* Clinical signs of pulmonary congestion, plus signs of impaired organ perfusion with at least one of the following manifestations:

  * altered mental status.
  * cold and clammy skin and limbs.
  * oliguria with a urine output of less than 30 ml per hour.
  * elevated arterial lactate level of >2.0 mmol per litre.

Exclusion Criteria:

* Any of the inclusion criteria not met and:

  1. Unwilling to provide informed consent.
  2. Echocardiographic evidence (recorded within 90 mins of end of PCI procedure) of mechanical cause for CS: eg ventricular septal defect, LV-free wall rupture, ischaemic mitral regurgitation.
  3. Age <18 and ≥80 years.
  4. Shock from another cause (sepsis, haemorrhagic/hypovolaemic shock, anaphylaxis, etc).
  5. Significant systemic illness
  6. Known dementia of any severity
  7. Comorbidity with life expectancy <12 months.
  8. Out-of-hospital cardiac arrest (OHCA) and any of the following:

     1. No return of spontaneous circulation (ongoing resuscitation effort)
     2. pH <7
     3. Without bystander CPR within 10 minutes of collapse
  9. Arterial lactate level of <2.0 mmol per litre.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to recruiting sites who fulfil study inclusion criteria and have no exclusion, will be considered. The majority of patients will be present through the heart attack centres and pathways. Some patients will, however, develop cardiogenic shock (CS) during their admission. These patients will be recruited from the coronary care units, intensive care units or cardiology wards and will be identified by clinicians who will alert research staff.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary aim is to better understand the heterogeneity of the immune consequences and treatment responses in CS through identification of transcriptomic sub-phenotypes and their association with in-hospital mortality | through study completion, an average of 5 days
  This will be achieved through bloods sample collection, analysis and linked to the patient's clinical diagnosis and outcome.

SECONDARY OUTCOMES:
Identify transcriptomic (and chemokine/cytokine) signatures at presentation that elucidate the pathobiology of CS and examine their subsequent evolution. | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.
Correlate recently identified clinical phenotypes of CS with transcriptomic and inflammatory mediator signatures. | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.
Identify transcriptomic and chemokine/cytokine signatures at presentation that improve prognostic accuracy in patients with CS | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.
Investigate inter-individual heterogeneity in the dynamic transcriptomic response to CS through an eQTL mapping approach and identify context- specific regulatory genetic variants involving gene networks central to the pathogenesis of CS. | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.
Identity novel therapeutic targets that might modulate the dysfunctional immune response to CS - "drug discovery" | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.
Determine the extent to which the signatures and drivers of a dysfunctional immune response in CS are shared with other critical illness syndromes. | through study completion, an average of 5 days
  Bloods samples will be collected from patients during their hospital stay and corresponding analysis performed.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Proudfoot, Principal Investigator — Barts Heath NHS trust
Locations (1):
- Barts Health NHS trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maslove DM, Tang B, Shankar-Hari M, Lawler PR, Angus DC, Baillie JK, Baron RM, Bauer M, Buchman TG, Calfee CS, Dos Santos CC, Giamarellos-Bourboulis EJ, Gordon AC, Kellum JA, Knight JC, Leligdowicz A, McAuley DF, McLean AS, Menon DK, Meyer NJ, Moldawer LL, Reddy K, Reilly JP, Russell JA, Sevransky JE, Seymour CW, Shapiro NI, Singer M, Summers C, Sweeney TE, Thompson BT, van der Poll T, Venkatesh B, Walley KR, Walsh TS, Ware LB, Wong HR, Zador ZE, Marshall JC. Redefining critical illness. Nat Med. 2022 Jun;28(6):1141-1148. doi: 10.1038/s41591-022-01843-x. Epub 2022 Jun 17. PMID 35715504
- [Background] Davenport EE, Burnham KL, Radhakrishnan J, Humburg P, Hutton P, Mills TC, Rautanen A, Gordon AC, Garrard C, Hill AV, Hinds CJ, Knight JC. Genomic landscape of the individual host response and outcomes in sepsis: a prospective cohort study. Lancet Respir Med. 2016 Apr;4(4):259-71. doi: 10.1016/S2213-2600(16)00046-1. Epub 2016 Feb 23. PMID 26917434
- [Background] Toma A, Dos Santos C, Burzynska B, Gora M, Kiliszek M, Stickle N, Kirsten H, Kosyakovsky LB, Wang B, van Diepen S, Epelman S, Szekely Y, Marshall JC, Billia F, Lawler PR. Diversity in the Expressed Genomic Host Response to Myocardial Infarction. Circ Res. 2022 Jun 24;131(1):106-108. doi: 10.1161/CIRCRESAHA.121.318391. Epub 2022 May 9. No abstract available. PMID 35534922
- [Background] Cano-Gamez K, Burnham KL, Goh C, Allcock A, Malick ZH, Overend L, Kwok A, Smith DA, Peters-Sengers H, Antcliffe D; GAinS Investigators; McKechnie S, Scicluna BP, van der Poll T, Gordon AC, Hinds CJ, Davenport EE, Knight JC, Webster N, Galley H, Taylor J, Hall S, Addison J, Roughton S, Tennant H, Guleri A, Waddington N, Arawwawala D, Durcan J, Short A, Swan K, Williams S, Smolen S, Mitchell-Inwang C, Gordon T, Errington E, Templeton M, Venatesh P, Ward G, McCauley M, Baudouin S, Higham C, Soar J, Grier S, Hall E, Brett S, Kitson D, Wilson R, Mountford L, Moreno J, Hall P, Hewlett J, McKechnie S, Garrard C, Millo J, Young D, Hutton P, Parsons P, Smiths A, Faras-Arraya R, Soar J, Raymode P, Thompson J, Bowrey S, Kazembe S, Rich N, Andreou P, Hales D, Roberts E, Fletcher S, Rosbergen M, Glister G, Cuesta JM, Bion J, Millar J, Perry EJ, Willis H, Mitchell N, Ruel S, Carrera R, Wilde J, Nilson A, Lees S, Kapila A, Jacques N, Atkinson J, Brown A, Prowse H, Krige A, Bland M, Bullock L, Harrison D, Mills G, Humphreys J, Armitage K, Laha S, Baldwin J, Walsh A, Doherty N, Drage S, Ortiz-Ruiz de Gordoa L, Lowes S, Higham C, Walsh H, Calder V, Swan C, Payne H, Higgins D, Andrews S, Mappleback S, Hind C, Garrard C, Watson D, McLees E, Purdy A, Stotz M, Ochelli-Okpue A, Bonner S, Whitehead I, Hugil K, Goodridge V, Cawthor L, Kuper M, Pahary S, Bellingan G, Marshall R, Montgomery H, Ryu JH, Bercades G, Boluda S, Bentley A, Mccalman K, Jefferies F, Knight J, Davenport E, Burnham K, Maugeri N, Radhakrishnan J, Mi Y, Allcock A, Goh C. An immune dysfunction score for stratification of patients with acute infection based on whole-blood gene expression. Sci Transl Med. 2022 Nov 2;14(669):eabq4433. doi: 10.1126/scitranslmed.abq4433. Epub 2022 Nov 2. PMID 36322631